CLINICAL TRIAL: NCT03124056
Title: Clinical and Biological Study of the Efficacy of the Use of Closed Extracorporeal Photopheresis in Acute or Chronic Graft Versus Host Disease After Allogeneic Hematopoietic Transplantation
Brief Title: Clinical and Biomarker Study of the Efficacy of Extracorporeal Photopheresis in Graft-versus-host Disease
Acronym: BIOECP_GVHD
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: 12/225
Record Dates: First submitted 2017-04-03; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Graft-versus-host Disease
Keywords: Extracorporeal photopheresis; Biomarker of response; Steroid resistant
MeSH Terms: conditions — Graft vs Host Disease | interventions — Photopheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Extracorporeal photopheresis — Extracorporeal photopheresis using non-open system

SUMMARY:
The aims of the study:

1. To evaluate the clinical efficacy of the use of extracorporeal photopheresis in the treatment of Graft-versus-host disease under standard clinical indications as pre-defined by the participants Centers (members of the Spanish Group for Hematopoietic Transplantation).
2. To explore and identify biomarkers of clinical response to extracorporeal photopheresis treatment of acute or chronic Graft-versus-host disease after Allogeneic hematopoietic stem cell transplantation

DETAILED DESCRIPTION:
Title: Exploratory study of biomarkers associated with clinical response to extracorporeal photopheresis in the treatment of acute and chronic graft-versus-host disease post allogeneic hematopoietic stem cell transplantation

Objectives:

1. To evaluate the clinical efficacy of the use of extracorporeal photopheresis in the treatment of acute or chronic Graft-versus-host disease under standard clinical indications as pre-defined by the participants Centers (Spanish Group for Hematopoietic Transplantation).
2. To explore and identify biomarkers of clinical response to extracorporeal photopheresis by means of a comprehensive analysis of different immune populations including T, B and Natural Killer cells, prior to and within the episodes of clinical graft-versus-host disease and the kinetic profile of plasma cytokines (Interferon-gamma, B cell activating factor, Tumor Necrosis Factor-alfa and Interleukin-6) in relation with Graft-versus-host disease .

Methods:

50 patients with acute or chronic graft-versus-host disease after Allogeneic hematopoietic stem cell transplantation whatever be the cell source (blood, bone marrow or cord blood), diagnosed and treated in one of the participant centers with closed extracorporeal photopheresis in the indications detailed bellow, will be analyzed in order to identify potential biomarkers of Graft versus host disease-response. Analyses of T, B and Natural Killer populations will be performed by Intracellular Cytokine Staining and Flow Cytometry. Cytokine measurement in plasma will be performed by Enzyme-Linked ImmunoSorbent Assay. Participants Centers:

* Hospital Clinico. Valencia. Spain
* Hospital Clinico. Salamanca. Spain
* Hospital Ramon y Cajal. Madrid. Spain.
* Hospital Murcia. Spain
* Hospital de Navarra, Pamplona. Spain

Each Centre will obtain approval of the study by the Local Ethical Committee and patients will sing inform consent. No risks are expected of the participation of the patients in this exploratory analytical study.

Frequency of treatment The frequency of treatment will depend on the type of Graft-versus-host disease (acute or chronic) and will be modified depending on the clinical response. All samples will be obtain at the same time that other standard blood samples.

Acute graft versus host disease: treatment will be initiated using 3 sessions/week, 1st week. Usually response will be determined in 3-4 weeks. If clear progression after 2 weeks of treatment or no response after 6-8 weeks treatment will be withhold and additional treatment will depend on the investigator decision. If response, the frequency of treatment will be reduced according to the following schedule:

* 2 treatments every week from week 2 to week 12
* 1 treatment every 2 weeks from week 13, until total suppression of corticosteroid treatment.

Response evaluation:

1. Complete remission: resolution of all signs of Graft-versus-host disease
2. Partial remission: improvement in at least 1 grade.
3. Absence of response

Chronic Graft-versus-host disease : treatment will be initiated using 3 sessions during week 1, 2 sessions every 2 weeks during weeks 2 to 12. If no progression, first evaluation will be done at 3 months (week 12). If no response, extracorporeal photopheresis will be withhold, except for sclerodermiform graft versus host disease in which evaluation will be done at 6 months. If response on week 12: 2 sessions every month for 3 additional months, after suppression of corticosteroid treatment. Use of NIH Consensus Group criteria of response (2006)

Biomarkers study: Samples: 2 x 10 ml whole blood in ethylenediaminetetraacetate. will be obtain in each time point analysis: pre-extracorporeal photopheresis and on days +7, +14, +21, +30 post-extracorporeal photopheresis in acute GVHD and pre-extracorporeal photopheresis and on days +15, +30, +45, +60, +75, +90 post-extracorporeal photopheresis in chronic Graft versus host disease. Samples will be processed in each participant Center in order to obtain mononuclear cells following the attached protocol and stored freezed until transportation to the Centralized processing Laboratory at the Hospital Clinico, Valencia, Spain and sending the clinical information included in the attached Excel Database.

1. Analyses of T, B and Natural Killer populations including Treg cells and dendritic cells Will be performed by Intracellular Cytokine Staining and Flow Cytometry (BD and Bioscience).

   Cell-populations and time-point to be monitored: pre-extracorporeal photopheresis and on days +7, +14, +21, +30 post-extracorporeal photopheresis in acute Graft versus host disease and pre-extracorporeal photopheresis and on days +15, +30, +45, +60, +75, +90 post-extracorporeal photopheresis in chronic Graft versus host disease.
2. Cytokine measurement in plasma (Interferon-gamma, Tumor Necrosis Factor-alfa, Interleukin-10, B cell activating factor and Interleukin-6)

ELIGIBILITY:
Inclusion Criteria:

Patients with acute or chronic graft-versus-host disease resistant or dependent to corticosteroids after Allogeneic Hematopoietic transplantation whatever be the cell source (blood, bone marrow or cord blood), diagnosed and treated in one of the participant centers

* Definitions:

Acute Graft versus host disease:

1. Refractory to corticosteroids: progression after 3-4 days of standard first line treatment with calcineurin inhibitor and glucocorticoids or no response after 7 days.
2. Corticosteroids dependent: flare o evidence of progression of Graft versus host disease in the same or new affected organ after reduction of full dose (2 mg/Kg/día), that has been maintained for at least 2 weeks.
3. Acute Graft versus host disease grade ≥ II, with response to 1st line treatment with cyclosporine A and prednisone in patients who present intolerable adverse effects that preclude to maintain this treatment as evaluated by the responsable physician.
4. Patient with viral reactivation during acute Graft versus host disease that need reduction of immunosuppression as evaluated by the responsable physician.

Chronic Graft versus host disease: Muco-cutaneous or hepatic moderate or severe chronic Graft versus host disease (as defined by NIH Consensus Group criteria (Biol Blood Marrow Transplantation 2005;11:945), refractory to steroids (1 mg/Kg/day of methylprednisolone during 15-30 days) or steroid-dependent (requiring more than 10 mg/day of methylprednisolone to control manifestations).

First line

* Associated to corticosteroids if exists contraindication for calcineurin inhibitors.
* Associated to calcineurin inhibitors and corticosteroids in case of pulmonary chronic Graft versus host disease diagnosis (optional) Second line
* Progressive cutaneous moderate or severe chronic Graft versus host disease after acute Graft versus host disease that is being treated with calcineurin inhibitors and corticosteroids.
* Moderate or severe cutaneous (both lichenoid or sclerodermiform) o mucosal chronic Graft versus host disease refractory to corticosteroids:

  * No Partial remission after 1 month of treatment
  * No Complete remission after 3 months of treatment
  * Disease progression after 2-3 weeks of treatment

Exclusion Criteria:

* uncontrolled Infections
* Performance score <3
* Lack of adequate vascular access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute or chronic graft-versus-host disease resistant or dependent to corticosteroids after Allogeneic hematopoietic stem cell transplantation whatever be the cell source (blood, bone marrow or cord blood), diagnosed and treated in one of the participant centers
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Graft versus host disease Response | 2 years
  Rate of clinical partial and complete response of acute and chronic Graft versus host disease to the intervention

SECONDARY OUTCOMES:
To determine rate of moderate and severe toxicity associated to extracorporeal photopheresis | 2 years
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0, Change From Baseline
To identify biomarkers associated with clinical response to extracorporeal photopheresis | 2 years
  Association between levels of peripheral blood lymphocyte populations or serum cytokines and Clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Solano, MD, PhD, Principal Investigator — Hospital Clinico of Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided